CLINICAL TRIAL: NCT03922217
Title: A Clinical Trial to Assess the Effect of Internet-delivered Mindfulness on Depressive Symptoms and Cognitive Function in Older Adults With Major Depression
Brief Title: e-Mindfulness for Depression in Older Adults
Acronym: MMW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201811036
Record Dates: First submitted 2019-03-13; First posted 2019-04-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Depression; Mental Health Disorder
MeSH Terms: conditions — Depression; Mental Disorders

STUDY DESIGN:
Intervention Model Description: open label
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental): This group will be given the Mindfulness mobile intervention, Mindful My Way (MMW)
  Interventions: Behavioral: Mindful My Way

INTERVENTIONS:
Behavioral: Mindful My Way — Mindful My Way (MMW) is a mobile application created for iOS, designed to delivered a form of mindfulness-based therapy to depressed older adults
  Other Names: MMW

SUMMARY:
This pilot study will test whether depression symptoms and cognitive functioning are impacted by internet-delivered mindfulness training following the principles of mindfulness meditation. The population is adults ages 65+ experiencing a current major depressive episode. Participants will receive an approximate 10-week instruction in mindfulness meditation, provided remotely through internet. Outcomes are depressive symptoms, assessed via clinical interview and self-report, and cognitive function, assessed via smartphone-delivered cognitive tests and surveys. The total duration of participation is approximately 18 weeks.

DETAILED DESCRIPTION:
The investigators will conduct a clinical trial using a smartphone app to collect data on depressive symptoms and cognitive function, and a website to deliver pre-recorded mindfulness sessions. The clinical trial will evaluate feasibility, acceptability, and efficacy with respect to depressive and cognitive symptoms, in a population of older adults at least 65 years of age with a current, active major depressive episode. This online, internet-delivered mindfulness meditation course is termed "Mindful My Way", consisting of 10 approximately one-hour classes consisting of mindfulness content (e.g., meditations) that a participant can watch on his or her computer or mobile device.

Assessment measures include a baseline diagnostic and screening assessment conducted by phone or RedCap survey, plus:

* Pre-mindfulness and post-mindfulness : (a) (1) 4 weeks of cognitive testing delivered via app (brief game-like tests delivered up to 4 times daily); and (2) 4 weeks of depressive symptom surveys (8 depressive symptoms delivered 4 times daily) end of study, (b) a MADRS via phone interview (brief clinical interview of depressive symptom severity).
* During the mindfulness class: questions on participant preferences in order to evaluate the feasibility and acceptability of the mindfulness course, delivered via app.

All of these remote smartphone-based assessment techniques have been previously used in Wash U IRB-approved studies. (IRB # 201612089, IRB # 201709118).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65 or older
* DSM-V diagnosis of Major Depressive Disorder or Bipolar, Depressed type and experiencing depressive symptoms consistent with current major depressive episode
* Not currently psychotic and no history of psychosis within the previous 12 months; psychosis reported in the distant past may not be exclusionary if brief, per PI's judgment
* English speaking
* Able to give informed consent
* iOS smartphone user with internet access
* iOS operating system 6 or newer
* Internet access to view internet mindfulness course

Exclusion Criteria:

* Confirmed psychotic disorder, history of primary post-traumatic stress disorder
* Current or recent substance use disorder that according to the PI's judgement would confound the interpretation of the study results
* Any severe Axis II personality disorder or psychotic disorder that, in the PI's judgement, could confound diagnosis or adherence to treatment
* Meets DSM-V criteria for Mental Retardation
* Acutely suicidal or homicidal (i.e., in imminent danger with plan, urges and intent to harm oneself or others including any prior serious attempts (e.g., those requiring hospitalization) at the PI discretion
* Current incarceration
* Inability to cognitively manage the tasks required in this study
* Unstable medical condition (e.g. uncontrolled diabetes mellitus or hypertension)
* Concurrent cognitive training, such as brain-training software, regular engagement in mindfulness practice and/or yoga x) significant neurological condition (e.g. stroke, seizure disorder, multiple sclerosis), that in the PI's judgment, could confound the interpretation of study results

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
EMA Depression Scale | Change from baseline, established during the 4 weeks preceding the intervention, which will be measured in the 4 weeks following completion of the intervention
  Scale Range: 0-8 (0-no depressive symptoms; 8-worst depressive symptoms measurable with this scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, Health Mind Lab, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schweiger A, Rodebaugh TL, Lenze EJ, Keenoy K, Hassenstab J, Kloeckner J, Gettinger TR, Nicol GE. Mindfulness Training for Depressed Older Adults Using Smartphone Technology: Protocol for a Fully Remote Precision Clinical Trial. JMIR Res Protoc. 2022 Oct 27;11(10):e39233. doi: 10.2196/39233. PMID 36301604